CLINICAL TRIAL: NCT01092338
Title: Safe and Effective Vitamin D Supplementation in HIV
Brief Title: Vitamin D Dose Finding Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-007332; R01AT005531 (NIH)
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Results first posted 2013-09-18 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-08

CONDITIONS: HIV Infections; AIDS
Keywords: Human Immunodeficiency Virus; Acquired Immune Deficiency Syndrome; Vitamin D; HIV; Complementary therapies
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 4000IU (Active Comparator): Subjects in this arm take a daily dose of 4000IU of Vitamin D3
  Interventions: Drug: Cholecalciferol (Vit D3)
- 7000IU (Active Comparator): Subjects in this arm of the study take a daily dose of 7000IU of Vitamin D3
  Interventions: Drug: Cholecalciferol (Vit D3)

INTERVENTIONS:
Drug: Cholecalciferol (Vit D3) — To test two oral daily doses (4000 vs. 7000 IU) of cholecalciferol (D3) dietary supplement (capsules or liquid) over a 3-month period in 44 children, adolescents and adults with HIV/AIDS.
  Other Names: Carlson D Drops: The D Drop Company; Nutraceutical Life Sciences Vitamin D3 2000 IU capsules: Vitacost; NOW Foods 5000 IU softgels: Now Health Group, Inc.

SUMMARY:
Optimal vitamin D (vit D) concentration and metabolism are essential for normal immune function, growth, muscle, bone, and inflammatory status in children, adolescents and adults with HIV/AIDS. The impact of vit D supplementation will be evaluated for safety and efficacy using clinically important outcomes, and this will overcome the critical barrier for use of vit D supplementation in research and clinical care. Inexpensive and easy to administer, vit D supplementation may prove to be an effective and feasible treatment for symptoms and prevention of side effects for people of all ages living with HIV/AIDS in the US and around the world.

DETAILED DESCRIPTION:
The key role of vitamin D (vit D) in maintaining optimal bone health has long been recognized, but its role in modulating the innate immune response and inflammatory reaction has only recently come under active investigation. As such, vit D is an increasingly frequently chosen and prescribed high dose dietary supplement,because it is thought to improve immune and inflammatory status in healthy people of all ages, and in those with chronic diseases including HIV/AIDS. Vit D also has calciotrophic functions essential for bone health, and poor vit D status contributes to the osteopenia/osteoporosis associated with antiretroviral therapy (ART). Vit D may improve insulin/glucose/lipid metabolism, blood pressure and risk of some cancers, all of which may complicate HIV/AIDS and its treatments. Poor vit D status is common in patients with HIV/AIDS of all ages and factors such as age, skin pigment, lactose intolerance and sun exposure alter the risks for vit D deficiency. In the multicenter U.S. REACH study of adolescents (72% African American), with and without HIV, showed that 87% had low serum 25D concentrations (<15 ng/mL), compared to 34% in a recent sample of healthy African American children from Philadelphia. Young African Americans are disproportionately affected by HIV infection in the US (~ 55% among persons with HIV aged 13 to 24 years are African American), and are also at high risk for vit D deficiency. Vit D therapy has great promise to improve major medical conditions and the quality of life for our patients with HIV/AIDS, yet the potential role of vit D in the treatment of HIV/AIDS has not been formally tested. Well-designed randomized trials are urgently needed to determine vit D supplementation safety and efficacy.

The investigators propose a two-phase study to establish safety and efficacy of high dose vit D supplementation in children and adults with HIV/AIDS. In Study Phase I, the safety and efficacy of two oral vit D3 doses (4000 and 7000 IU/d) are determined over 12 weeks in 44 subjects ages 5.0 to 24.9 y. The key safety measure is concurrently elevated serum calcium and 25D concentrations. Efficacy is evaluated by serum 25D concentration and cathelicidin (innate immune, antimicrobial protein) mRNA expression. Study Phase II is a 12 month, double blind, randomized, placebo controlled supplementation study (n=52). Key outcomes include safety and longterm 25D concentration within the goal range (32 to 160 ng/mL), improved cathelicidin mRNA expression, and measures of bone, muscle, inflammation, growth and body composition status, and HIV/AIDS disease severity. Based on the evidence and promise, vit D clearly deserves to be among the first nutrients evaluated in the National Center for Complimentary and Alternative Medicine (NCCAM) HIV research program.

ELIGIBILITY:
Inclusion Criteria:

1. HIV seropositive diagnosed with standard techniques
2. Age for perinatally-acquired HIV/AIDS Group (PA subjects): 5.0 to 24.9 y
3. Age for non-perinatally-acquired HIV/AIDS Group (non-PA subjects): 15.0 to 24.9 y
4. In usual state of good health (no hospitalizations, emergency room or unscheduled acute illness visits for 2 weeks prior)
5. Subject and/or family commitment to the 3-month study

Exclusion Criteria:

1. Other chronic health conditions that may affect growth, dietary intake, and/or nutritional status
2. Pregnancy
3. Participation in another HIV intervention study with impact on 25D serum concentrations
4. Use of vit D supplementation (subjects willing to discontinue supplementation will become eligible after a 2-month washout period)
5. Baseline elevated serum calcium concentration
6. Non-English speaking

Ages: 5 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Stallings, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Groleau V, Herold RA, Schall JI, Wagner JL, Dougherty KA, Zemel BS, Rutstein RM, Stallings VA. Blood lead concentration is not altered by high-dose vitamin D supplementation in children and young adults with HIV. J Pediatr Gastroenterol Nutr. 2013 Mar;56(3):316-9. doi: 10.1097/MPG.0b013e3182758c4a. PMID 23059649
- [Derived] Dougherty KA, Schall JI, Zemel BS, Tuluc F, Hou X, Rutstein RM, Stallings VA. Safety and Efficacy of High-Dose Daily Vitamin D3 Supplementation in Children and Young Adults Infected With Human Immunodeficiency Virus. J Pediatric Infect Dis Soc. 2014 Dec;3(4):294-303. doi: 10.1093/jpids/piu012. Epub 2014 Mar 27. PMID 26625449

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Study started enrollment in 01/2010 and completed in 01/2011. A total of 44 subjects were enrolled including 19 with perinatally-acquired HIV/AIDS (PA) and 25 with behaviorally-acquired HIV/AIDS (BA).
Pre-assignment Details: Subjects taking a vitamin D supplement or multi-vitamin were eligible if they were willing to discontinue supplementation after a minimum of a 2 month washout period.
Period: Overall Study
Arm/Group | 4000IU/d of Vitamin D3 | 7000IU/d Vitamin D3
Started | 22 | 22
Completed | 21 | 21
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4000IU/d of Vitamin D3 | 7000IU/d Vitamin D3 | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 7 | 16
  Between 18 and 65 years | 13 | 15 | 28
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 18.4 (4.5) | 19.1 (5.0) | 18.7 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 15 | 15 | 30
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Safety
Description: Determined by incidence of elevated serum calcium (above age specific range) associated with elevated serum 25D concentrations (>160ng/ml).
Time Frame: 12 weeks
Population: Number of subjects with elevated serum calcium (above age specific range) associated with elevated serum 25D concentrations (>160ng/ml)
Measure: Number; unit: participants
Arm/Group | 4000IU/d of Vitamin D3 | 7000IU/d Vitamin D3
Number analyzed (Participants) | 22 | 22
participants | 0 | 0

2. Primary Outcome: Efficacy of the Two Doses (4000 and 7000 IU/d)
Description: Daily D3 supplementation will result in 25D >= to 32/ng/ml
Time Frame: 12 weeks
Population: Number of subjects with serum 25D concentration levels >= 32 ng/ml after 12 weeks of supplementation.
Measure: Number; unit: participants
Arm/Group | 4000IU/d of Vitamin D3 | 7000IU/d Vitamin D3
Number analyzed (Participants) | 22 | 22
participants | 16 | 19

ADVERSE EVENTS:
Arm/Group | 4000IU/d of Vitamin D3 | 7000IU/d Vitamin D3
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 12/22 | 10/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4000IU/d of Vitamin D3 (N=22) | 7000IU/d Vitamin D3 (N=22)
nausea (Gastrointestinal disorders) | 3 (3) | 4 (5)
General (General disorders) | 4 (5) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Infection (Infections and infestations) | 4 (4) | 1 (2)
Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Cough/Cold (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No